CLINICAL TRIAL: NCT03794830
Title: The Influence of the Manipulation of the Sacroiliac Joint on Low Back Pain With or Without Radiation to Lower Limbs
Brief Title: The Influence of the Manipulation of the Sacroiliac Joint on Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Alejandro Caña Pino, Principal Investigator. Medical Surgical-Therapy Department, Universidad de Extremadura Facultad de Medicina, Badajoz, Spain, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 041218
Record Dates: First submitted 2019-01-03; First posted 2019-01-07 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Low Back Pain; Sacroiliac Disorder
Keywords: sacroiliac joint; low back pain; Osteopathic manipulation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manipulation group (MG) (Experimental): Patients were treated with sacroiliac joint osteopathic semidirect manipulation twice a week every 3 to 4 days over a period of time of 3 weeks
  Interventions: Other: manipulation group (MG)
- electrotherapy group (EG) (Active Comparator): Patients were treated with micro-waves (circular antenna in lumbar area, pulsating-mode 120W for 12 minutes) and later conventional analgesic TENS (80Hz frequency, 30 minutes) 5 days per week over a period of time of 3 weeks (15 sessions of electrotherapy).
  Interventions: Other: electrotheraphy group (EG)

INTERVENTIONS:
Other: manipulation group (MG) — Patients were treated with sacroiliac joint osteopathic semidirect manipulation twice a week every 3 to 4 days over a period of time of 3 weeks
  Arms: manipulation group (MG)
Other: electrotheraphy group (EG) — Patients were treated with micro-waves (circular antenna in lumbar area, pulsating-mode 120W for 12 minutes) and later conventional analgesic TENS (80Hz frequency, 30 minutes) 5 days per week over a period of time of 3 weeks (15 sessions)
  Arms: electrotherapy group (EG)

SUMMARY:
The primary focus of this study is to know the influence of sacroiliac joint manipulation on low back pain with or without radiation to lower limbs, in the lumbopelvic-hip joint

DETAILED DESCRIPTION:
One of the main problems faced by physiotherapists in primary care is low back pain with or without radiation to lower limbs. Nowadays, there are a lot of types of low back pain interventions, yet despite the vast amount of research findings, the evidence remains contradictory and inconclusive: Pharmacological treatments like NSAIDs have shown result in acute low back pain but not in chronic pain; conservative interventions (ultrasound, interferential currents, mechanical traction and massage) have been studied and found ineffective.

A total of 151 low back pain patients with or without radiation to lower limbs between 18-70 years old derived from the Physiotherapy Unit of Gévora Health Center (Badajoz, Spain) voluntarily entered the study

ELIGIBILITY:
Inclusion Criteria:

* dysfunction or sacroiliac joint hypomobility (SI)
* having stopped taking anti-inflammatory medicines or analgesics three days before the study began

Exclusion Criteria:

* destructive injuries of the spine and pelvis
* fractures
* lumbar surgery
* sacroiliac instability
* spondylolisthesis
* pregnancy in progress
* cauda equina syndrome
* abdominal aneurysm
* infection
* inflammatory arthritis
* tumors
* osteoporosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-01-04 (Actual)

PRIMARY OUTCOMES:
visual analogue scale (VAS) | 1 week
  Pain assessment from 0 to 10. 0: no pain 10: maximum pain
Oswestry disability index (ODI) | 1 week
  disability assessment 0% -20% (Minimum Disability) 21% -40% (Moderate disability) 41% -60% (Severe disability) 61% -100% (Disabled):
Roland Morris questionnaire | 1 week
  disability assessment The extreme values oscillate between 0 (absence of disability due to low back pain) and 24 (maximum possible disability)
digital algometer (Wagner, FPIX model) | 1 week
  Pain threshold assessment by pressing the sensitive points of the muscle

CONTACTS AND LOCATIONS:
Overall Officials: Jose Antonio JA Rodriguez-Pastor, PhD, Principal Investigator — Universidad de Extremadura. Facultad de Medicina (Badajoz). Spain; Mª Dolores MD Apolo-Arenas, PhD, Study Director — Universidad de Extremadura. Facultad de Medicina (Badajoz). Spain; Berta BC Caro-Puértolas, PhD, Study Director — Universidad de Extremadura. Facultad de Medicina (Badajoz). Spain; Alejandro AC Caña-Pino, PT,MSc, Principal Investigator — Universidad de Extremadura. Facultad de Medicina (Badajoz). Spain
Locations (1):
- Universidad de Extremadura, Badajoz, Spain